CLINICAL TRIAL: NCT04826133
Title: Testing Restoring Effects of Vitamin D on the Dopamine System: A Human Laboratory Study Among Cocaine Users.
Brief Title: Vitamin D and Cocaine Administration
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Could not obtain additional funding to continue the research.
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Marc Potenza, Principal Investigator, Yale University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2000025367
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acute Pretreatment with Calcitriol (Active Comparator): To explore the effects of acute pre-treatment with Calcitriol on attempts to self-administer and ultimate number of infusions/boluses of cocaine, in experienced, non treatment-seeking users of the drug
  Interventions: Drug: Calcitriol
- Acute Pretreatment with Placebo (Placebo Comparator): To explore the effects of acute pre-treatment with placebo on attempts to self-administer and ultimate number of infusions/boluses of cocaine, in experienced, non treatment-seeking users of the drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calcitriol — Subjects will receive an oral administration of calcitriol (1,25-dihydroxyvitamin D3) 1.5 μg (three capsules of 0.5 μg each) at 9 pm, night before each cocaine session, and at 8 am, morning of each cocaine session. This dose of calcitriol is lower than doses safely administered in other human studies and for a duration of time shorter than doses safely administered in other trials. In addition, this dose has been already tested by our group, subject of a different grant application, and should be effective at enhancing stimulant's induced dopamine release, in comparison to placebo.
  Other Names: 1,25-dihydroxyvitamin D3
  Arms: Acute Pretreatment with Calcitriol
Other: Placebo — Subjects will receive an oral administration of three capsules of placebo at 9 pm the night before each cocaine session, and at 8 am, morning of each cocaine session.
  Arms: Acute Pretreatment with Placebo

SUMMARY:
This study is designed to explore the effects of acute pre-treatment with 1,25-dihydroxyvitamin D3 (calcitriol), as compared to placebo on the behavioral (e.g., attempts to self-administer and ultimate number of infusions/boluses of cocaine self-administered), neurocognitive (e.g., performance on computerized tests of reward related learning such as the probabilistic selection task or PST and probabilistic reward task or PRT), and subjective effects (e.g, computerized visual analog scale [VAS] ratings of euphoria/, craving, etc.) of cocaine in experienced, non-treatment seeking users of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-55 years
* Voluntary, written, informed consent
* Physically healthy by medical history, physical, neurological, ECG and laboratory examinations
* DSM-5 criteria for at least moderate Cocaine Use Disorder
* Recent street cocaine use in excess of quantities used in the current study
* Intravenous and/or smoked (crack/ freebase) use
* Positive urine toxicology screen for cocaine
* Laboratory evidence of vitamin D sufficiency (i.e., 25(OH)-vitamin D3 level ≥ 20/mg)
* For females, a negative serum pregnancy (HCG) test at screening and admission, and a negative urine pregnancy test (HCG) on cocaine administration days.

Exclusion Criteria:

* A history of other substance dependence (except for nicotine). Positive urine toxicology for cannabis is accepted for the study unless there is evidence for dependence per Structured Clinical Interview for DSM-5 (SCID) interview. Positive urine toxicology for other drugs at screening will be repeated. If positive again and/or positive at admission, subjects will be excluded
* < 1 year of cocaine abuse/dependence
* A primary DSM-5 Axis I major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) unrelated to cocaine as determined by the SCID-5
* Medical comorbidities including serum calcium ( > 10.5 mg/dl, serum phosphorus > 4.2 mg/dl), hyperparathyroidism, kidney disease (e.g., Serum creatinine > 1.3 mg/dl)
* A history of significant and uncontrolled medical (e.g., cardiovascular, diabetic/metabolic) or neurological (e.g., cerebrovascular, seizures, traumatic brain injury) illness
* A history of seizures
* Current use of psychotropic/potentially psychoactive medications or medications that can have drug drug interactions with calcitriol, including over the counter Vitamin D products, thiazide diuretics, and calcium supplements, etc, as referenced in the package insert for calcitriol
* Seeking treatment for drug abuse/dependence
* Hypersensitivity to calcitriol
* For females, physical or laboratory (HCG) evidence of pregnancy.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Cocaine Self Administration Attempts | 90 minutes
  Number of attempts to self administer cocaine will be analyzed.
Cocaine Self Administration Infusions | 90 minutes
  Number of infusions of cocaine will be analyzed.

SECONDARY OUTCOMES:
Probabilistic Selection Task (PST) | 15 minutes
  The Probabilistic Selection Task (PST) is a computerized task that assesses the tendency to learn from positive versus negative outcomes. PST will be analyzed using linear mixed models with treatment and time included as a within subjects variable.
Probabilistic Reward Task (PRT) | 15 minutes
  The Probabilistic Reward Task (PRT) is a computerized task that uses an asymmetric reinforcement schedule to produce a response bias towards the more frequently rewarded of two possible stimuli. PRT will be analyzed using linear mixed models with treatment and time included as a within subjects variable.
Subjective Effects of Cocaine / Visual Analog Scale (VAS) | 150 minutes
  During cocaine sessions, subjects will complete a series of self rated subjective effects measuring how they feel on cocaine, using a scale of 0 (not at all) to 10 (most ever). VAS ratings will focus on euphoria ("high") as a primary outcome, however, other positive, negative, psychomotor, and drug-craving ratings (e.g. good, bad, stimulated, paranoid, hungry, etc.) will be collected as well. Ratings are implemented on a touch-screen laptop computer and presented every 5 minutes, throughout the session

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States